CLINICAL TRIAL: NCT07195526
Title: Getting Seniors Back on Their Bicycle; a Pretest-posttest Case-control Study on the Improvement of Bicycle Balance Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Responsible Party: Principal Investigator, Eric Maris, Principal Investigator, Donders Centre for Cognitive Neuroimaging
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCC.2024.00080
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Balance Control in Elderly
Keywords: Balance control; bicycle balance; motor skill training; mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bicycle balance control training (Experimental): The intervention involveds three components: (1) training on an exercise bicycle, (2) a balance control training on a bicycle simulator, and (3) cycling on the public roads with a safe start-and-stop technique that will be practiced on the bicycle simulator. In the bicycle simulator training, the difficulty of the balance control was increased gradually, slowly approaching the difficulty of bicycle balance control on the public roads.
  Interventions: Behavioral: Bicycle balance control training
- Control group (No Intervention): The participants in the experimental group are matched to the participants in the control group. The control group participants are selected based on their distance from the location of the intervention; control group participants live farther away from the location of the intervention as compared to the experimental group.

INTERVENTIONS:
Behavioral: Bicycle balance control training — The intervention involves three components: (1) training on an exercise bicycle, (2) a balance control training on a bicycle simulator, and (3) cycling on the public roads with a safe start-and-stop technique that was practiced on the bicycle simulator. In the bicycle simulator training, the difficulty of the balance control will be increased gradually, slowly approaching the difficulty of bicycle balance control on the public roads.
  Arms: Bicycle balance control training

SUMMARY:
This study investigates the effectiveness of an intervention that aims at restoring bicycle balance control skills in seniors that have quit cycling. The intervention will last 11 weeks and involves three components: (1) training on an exercise bicycle, (2) a balance control training on a bicycle simulator, and (3) cycling on the public roads with a safe start-and-stop technique that was practiced on the bicycle simulator. In the bicycle simulator training, the difficulty of the balance control will be increased gradually, slowly approaching the difficulty of bicycle balance control on the public roads.

ELIGIBILITY:
Inclusion Criteria:

* Persons that stopped cycling at least six months ago and want to get back on their bicycle.

Exclusion Criteria:

* Balance-relevant sensory disorders (peripheral neuropathy, labyrinthitis, vestibular neuritis, …)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Bicycle balance control skill and confidence | Pretest: Between the second and the third week of June 2023 Posttest: First week of October 2023
  This outcome variable will be obtained from a questionnaire that evaluates participants' bicycle BC skills and confidence while riding on the public roads. For each of three environments (without traffic, little traffic, busy traffic), participants must indicate what applies to them: (1) "I did not ride my bicycle here", (2) "I rode my bicycle here, but I try to avoid it", and (3) "I rode my bicycle here without problems". The answers to every question/environment were converted into a score by assigning 0, 1, and 2 points to the respective options. Summing these scores over the three questions/environments results in a number between 0 and 6, which is the outcome variable.

SECONDARY OUTCOMES:
One-minute functional threshold power (1minFTP) | From the third week of June 2023 until the second week of August 2023
  The 1minFTP is the highest power a participant can maintain for one minute while cycling at 60 revolutions per minute (RPM). The 1minFTP was assessed by having participants monitor their breath after a one-minute effort at some power level: if the participant can say only a few words at a time (a proxy for reaching the ventilatory threshold), the 1minFTP is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Maris, PhD, Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (1):
- Faculty of Social Sciences Research labs and Radboud University Sports Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT07195526/ICF_000.pdf